CLINICAL TRIAL: NCT02310243
Title: Phase Ib/IIa Study of Palbociclib in MLL-rearranged Acute Leukemias AMLSG 23-14/Palbo-AL-1
Brief Title: Study of Palbociclib in MLL-rearranged Acute Leukemias
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Ulm (Other)
Collaborators: Pfizer (Industry); National Center for Tumor Diseases, Heidelberg (Other)
Responsible Party: Principal Investigator, Peter Paschka, Prof. Dr. med., University of Ulm
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMLSG 23-14
Record Dates: First submitted 2014-12-01; First posted 2014-12-08 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia
Keywords: Acute myeloid leukemia; Acute lymphoblastic leukemia; MLL-rearranged leukemia; Palbociclib (PD-0332991-00)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Palbociclib (Experimental): Phase1b: 125 mg palbociclib once daily for 21 days followed by 7 days of rest; this regimen will be chosen for the first dose to be evaluated.
  phase IIa: single-agent palbociclib using the tolerable dose defined in the phase Ib part of the study is administered once daily for 21 days followed by 7 days of rest.
  Interventions: Drug: Palbociclib

INTERVENTIONS:
Drug: Palbociclib — oral, once daily (125mg, 100mg or 75mg) for 21 days
  Other Names: PD-0332991-00

SUMMARY:
Diagnosis: Acute myeloid leukemia; Acute lymphoblastic leukemia Age ≥ 18 years, no upper age limit Study drug: Palbociclib Phase Ib/IIa, open-label

* Phase Ib: Based on previous experience with 125 mg palbociclib once daily for 21 days followed by 7 days of rest in patients with breast cancer, liposarcoma, non-small cell lung cancer, hepatocellular carcinoma, ovarian cancer, mantle-cell lymphoma, and glioblastoma, this regimen will be chosen for the first dose to be evaluated in the phase Ib. Based on a 3 + 3 modified Fibonacci design, the tolerable dose of palbociclib for the phase IIa is defined.
* Phase IIa: single-agent palbociclib using the tolerable dose defined in the phase Ib part of the study is administered once daily for 21 days followed by 7 days of rest. Based on the optimal two-stage design of Simon, 21 patients are treated in the first stage. If results are positive, 29 additional patients will be recruited into the second stage of the study. An efficacy of the investigational therapy will be rejected in the first stage of 21 treated patients if two or less patients achieve complete remission (CR), CR with incomplete blood count recovery (CRi), partial remission (PR), or anti-leukemic effect (ALE). If three or more patients achieve CR, CRi, PR, or ALE during this first stage, the trial is intended to be continued in the second stage with a total sample size of 50 patients.

Start of recruitment: July 2015 End of recruitment: July 2017 End of study (last patient out): July 2018 The treatment duration of an individual patient is estimated to be 2-6 months, but may be unlimited in patients with sustained response ("case-by-case decision").

Observation time per patient after entry into the study (incl. treatment) is at least 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed diagnosis of acute leukemia with MLL rearrangement according to the 2008 WHO Classification
* Patients with MLL-rearranged leukemia who are refractory to standard induction therapy and not immediate candidates for allogeneic HSCT (bridge to transplant is allowed)
* Patients with MLL-rearranged leukemia who relapsed after standard first-line treatment and are not immediate candidates for allogeneic HSCT (bridge to transplant is allowed)
* Patients with newly diagnosed MLL-rearranged leukemia who are not eligible for intensive first-line therapy
* Genetic/histologic/immunohistologic assessment in one of the central laboratories
* Age ≥ 18 years, no upper age limit
* WHO performance status of ≤ 2
* No prior chemotherapy two weeks before study entry except hydroxyurea to control hyperleukocytosis
* Non-pregnant and non-nursing. Women of child-bearing potential must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 72 hours prior to registration (WOCBP is defined as a sexually active mature woman who has not undergone a hysterectomy or who has had menses at any time in the preceding 24 months).
* Female patients in the reproductive age and male patients must agree to avoid getting pregnant or to father a child while on therapy and for three months after the last dose of therapy.
* Women of child-bearing potential must either commit to continued abstinence from heterosexual intercourse or begin one acceptable method of birth control (IUD, tubal ligation, or partner's vasectomy). Hormonal contraception is an inadequate method of birth control.
* Men must agree not to father a child and must use a latex condom during any sexual contact with WOCBP while receiving therapy and for three months after therapy is stopped, even if they have undergone successful vasectomy.
* Signed written informed consent

Exclusion Criteria:

* Prior treatment with palbociclib
* Performance status > 2 according to WHO criteria
* Organ insufficiency: creatinine > 1.5 x upper normal serum level; bilirubin, AST, or AP > 2.5 x upper normal serum level; heart failure NYHA III/IV; uncontrolled hypertension; unstable angina; serious cardiac arrhythmia; severe obstructive or restrictive ventilation disorder
* Uncontrolled infection
* Patients with a "currently active" second malignancy other than non-melanoma skin cancer. Patients are not considered to have a "currently active" malignancy if they have completed therapy and are considered by their physician to be at less than 30% risk of relapse within one year.
* Severe neurologic or psychiatric disorder interfering with ability of giving informed consent
* Known or suspected active alcohol or drug abuse
* Known positivity for HIV, active HAV, HBV, or HCV infection
* Bleeding disorder unrelated to leukemia
* Uncontrolled CNS involvement (treatment for CNS-involvement prior to inclusion is allowed)
* QTc > 470 msec (based on the mean value of triplicate ECGs), family or personal history of long or short QT syndrome, Brugada syndrome, or known history of QTc prolongation or Torsade de Pointes
* Uncontrolled electrolyte disorders that can aggravate the effects of a QTc-prolonging drug (e.g., hypocalcemia, hypokalemia, hypomagnesemia)
* No consent for registration, storage, and processing of individual disease characteristics, information on the course of the disease, and information obtained from the family physician and/or other physicians involved in the treatment of the patient about study participation
* No consent for biobanking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-07; Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | 12 months
  Safety assessments
Maximum tolerated dose of palbociclib | 12 months
overall response rate | 12 months

SECONDARY OUTCOMES:
Relapse-free survival | three years
Overall survival | three years
Evaluation of target (CDK6) inhibition by palbociclib | three years
Assessment of Quality of life | 6 months

CONTACTS AND LOCATIONS:
Locations (24):
- Germany (24):
  - Klinikum Augsburg, Augsburg
  - Helios Klinikum Bad Saarow, Bad Saarow
  - Charité Campus Benjamin Franklin, Berlin
  - Vivantes Klinikum Neukölln, Berlin
  - Charité Campus Virchow-Klinikum, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Städtisches Klinikum Braunschweig gGmbH, Braunschweig
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Kliniken Essen Süd, Ev. Krankenhaus Essen-Werden gGmbH, Essen
  - Malteser Krankenhaus St. Franziskus-Hospital, Flensburg
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - MVZ Osthessen, Fulda
  - Universitätsklinikum Giessen, Giessen
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - Städtisches Klinikum Karlsruhe gGmbH, Karlsruhe
  - Universitätsklinikum Schleswig-Holstein Campus Kiel, Kiel
  - Caritas-Krankenhaus Lebach, Lebach
  - Uni-Klinikum der Otto-von-Guericke-Universität, Magdeburg
  - Universitätsmedizin der Johannes Gutenberg-Universität, Mainz
  - Pius Hospital Oldenburg, Oldenburg
  - Medizinische Universitätsklinik Tübingen, Tübingen
  - University Hospital of Ulm, Ulm